CLINICAL TRIAL: NCT00665574
Title: A Prospective, Multi-center, Randomized, Double-blind Feasibility Study to Evaluate the Safety and Performance of ActaVisc and ActaVisc Mx Intra-articular Injection for Management of Pain Associated With Osteoarthritis in the Knee.
Brief Title: ActaVisc and ActaVisc Mx Intra-articular Injection for Pain Associated With Osteoarthritis in the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Carbylan Therapeutics, Inc. (Industry)
Responsible Party: Marcee Maroney, V.P. Marketing and Clinical Affairs, Carbylan BioSurgery, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIM 1.0
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ActaVisc
  Interventions: Other: ActaVisc and ActaVisc Mx Intra-articular Injection
- 2 (Experimental): ActaVisc Mx Intra-articular Injection
  Interventions: Other: ActaVisc and ActaVisc Mx Intra-articular Injection
- 3 (Placebo Comparator): Saline
  Interventions: Other: ActaVisc and ActaVisc Mx Intra-articular Injection
- 4 (Active Comparator): Corticosteroid
  Interventions: Other: ActaVisc and ActaVisc Mx Intra-articular Injection

INTERVENTIONS:
Other: ActaVisc and ActaVisc Mx Intra-articular Injection — ActaVisc is a hyaluronan based device intended to alleviate the pain associated with osteoarthritis of the knee with a single injection and ActaVisc Mx is the same material combined with a corticosteroid.

SUMMARY:
To evaluate the safety and performance of ActaVisc™ intra-articular injection (ActaVisc) and ActaVisc Mx, for management of pain associated with osteoarthritis in the knee in patients who have failed to respond adequately to conservative non-pharmacologic therapy and simple analgesics

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (OA) grade 2 or 3.
* Symptoms in the treatment knee for at least 12 months.
* Fully ambulatory patient.

Exclusion Criteria:

* Secondary OA resulting from rheumatoid arthritis, chondrocalcinosis, osteonecrosis, chronic fibromyalgia or other autoimmune disease.
* Generalized symptomatic OA in lower extremity joints other than the knees, inflammatory joint disease, bursitis, OA in the hips, or other condition that may interfere with study assessments.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the WOMAC Pain subscale average score for the treatment knee. | 26 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Latvia (2):
  - Daugavpils Pilsetas Centrala Slimnica, Daugavpils
  - State Hospital of Traumatology and Orthopaedics, Riga